CLINICAL TRIAL: NCT01771978
Title: Effects of Diltiazem and/or N-Acétylcystéine Versus Placebo on hémodynamiques and Biological Repercussions of the Ischaemia-réperfusion During the Coronary Surgery With Beating Heart
Brief Title: Ischaemia-réperfusion During the Coronary Surgery With Beating Heart
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2276
Record Dates: First submitted 2012-12-27; First posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2008-02

CONDITIONS: Ischaemia-reperfusion Injury
Keywords: ischaemia-reperfusion injury; cardiac surgery; oxidative stress markers; troponin; diltiazem; acetylcystein
MeSH Terms: conditions — Reperfusion Injury | interventions — Diltiazem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm1: control group (Placebo Comparator): Received 250 ml of a 5% dextrose solution as placebo drug
  Interventions: Drug: Placebo
- Arm 2: diltiazem group (Experimental): Received a 100 µg/kg bolus followed by a 0.3 µg/kg infusion diluted in 250 ml of 5% dextrose solution
  Interventions: Drug: Diltiazem
- Arm 3: acetylcystein group (Experimental): Received 150 mg/kg acetylcystein diluted in 250 ml of 5% dextrose solution
  Interventions: Drug: Acetylcystein
- Arm 4: diltiazem and acetylcystein group (Experimental): Received a combination of drug :
  bolus diltiazem 100 µg/kg followed by a 0.3 µg/kg infusion diluted in 125 ml of a 5% dextrose solution and 150 mg/kg acetylcystein diluted in 125 ml of 5% dextrose solution
  Interventions: Drug: diltiazem and acetylcystein

INTERVENTIONS:
Drug: Placebo — Received 250 ml of a 5% dextrose solution as placebo
  Other Names: placebo group
  Arms: Arm1: control group
Drug: Diltiazem — Received a 100 µg/kg bolus followed by a 0.3 µg/kg infusion diluted in 250 ml of 5% dextrose solution
  Other Names: Diltiazem group
  Arms: Arm 2: diltiazem group
Drug: Acetylcystein — Received 150 mg/kg acetylcystein diluted in 250 ml of 5% dextrose solution
  Other Names: Acetylcystein group
  Arms: Arm 3: acetylcystein group
Drug: diltiazem and acetylcystein — Received a combination of drug :diltiazem and acetylcystein
  * bolus diltiazem 100 µg/kg followed by a 0.3 µg/kg infusion diluted in 125 ml of a 5% dextrose solution
  * 150 mg/kg acetylcystein diluted in 125 ml of 5% dextrose solution
  Other Names: Combined diltiazem and acetylcystein drug group
  Arms: Arm 4: diltiazem and acetylcystein group

SUMMARY:
Less oxidative stress occurs during off-pump than on-pump coronary artery bypass graft (CABG) surgery but warm ischaemia-reperfusion injury may occur following transient coronary artery clamping. The aim of this study was to compare the preventive effects of diltiazem and N-acetylcysteine (NAC), alone or in combination, on biomarkers of myocardial damage and oxidative stress during off-pump CABG surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age included between 60 and 80 years

Exclusion Criteria:

* Age < 60 or > 80 years
* Pregnancy
* The allergy in used medicines (N-acétylcystéine, Diltiazem)
* Presence of a pathology valvulaire associated
* Urgency
* Unstable angor
* Bypass as a matter of urgency
* Recours peropératoire to a CEC
* FE < 0,40
* BAV of the 2nd and 3rd not sailed degree
* fibrillation or flutter little finger.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2002-06; Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Reduce the percentage 40% of patients operated on a beating heart to 10% as a result of treatment with diltiazem and N-acetylcysteine | during ischaemia-reperfusion
  Choosing as main biological variable rate cTnI cardiospecific, above the threshold of detection (0.3 mcg / L) in 40% of patients operated on a beating heart hoping to reduce this percentage to 10% as a result of treatment with diltiazem and N-acetylcysteine

CONTACTS AND LOCATIONS:
Overall Officials: Annick Steib, MD, PhD, Study Director — Strasbourg University Hospital, France
Locations (1):
- Department of Anaesthesiology, Strasbourg, France